CLINICAL TRIAL: NCT00898404
Title: Molecular Correlates of Methotrexate in Childhood ALL
Brief Title: Response or Resistance to Chemotherapy in Young Patients With Acute Lymphoblastic Leukemia Treated With Methotrexate
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL04B1; NCI-2009-00308 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000346452 (Other: Clinical Trials.gov); COG-AALL04B1 (Other: Children's Oncology Group); R01CA076641 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: B-cell Childhood Acute Lymphoblastic Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Recurrent Childhood Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm I: Tumor diagnostic specimens from patients who subsequently failed therapy within 4 years of diagnosis or who did not fail therapy within 4 years of diagnosis (control patients) are obtained from the Children's Oncology Group cellbank. Specimens are studied for molecular determinants of human reduced folate carrier (hRFC) gene expression and gene sequence alterations using reverse transcriptase-polymerase chain reaction (RT-PCR), thymidylate synthase inhibition assay, Rnase protection assay, or 5'RACE. Multidrug resistance proteins are also studied by RT-PCR.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is looking at response or resistance to chemotherapy in young patients with acute lymphoblastic leukemia treated with methotrexate. Studying samples of tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and drug resistance in patients.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the molecular basis for human reduced folate carrier (hRFC) transcripts in B-precursor and T-cell acute lymphoblastic leukemia (ALL) blasts obtained from children with newly diagnosed ALL subsequently treated with methotrexate.

II. Correlate hRFC expression in these specimens with methotrexate transport and sensitivities.

III. Determine the roles of high frequency gene/transcript variants for hRFC as determinants of response and resistance to methotrexate in these patients.

IV. Determine the roles of multidrug resistance-associated proteins as determinants of response and resistance to methotrexate and mercaptopurine in these patients.

OUTLINE: This is a multicenter study.

Tumor diagnostic specimens from patients who subsequently failed therapy within 4 years of diagnosis or who did not fail therapy within 4 years of diagnosis (control patients) are obtained from the Children's Oncology Group cellbank. Specimens are studied for molecular determinants of human reduced folate carrier (hRFC) gene expression and gene sequence alterations using reverse transcriptase-polymerase chain reaction (RT-PCR), thymidylate synthase inhibition assay, Rnase protection assay, or 5'RACE. Multidrug resistance proteins are also studied by RT-PCR.

A certificate of confidentiality protecting the identity of research participants in this project has been issued by the National Cancer Institute.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-precursor or T-cell acute lymphoblastic leukemia

  * Newly diagnosed disease subsequently treated with methotrexate
* Banked diagnostic blast specimens are available from Childrens Oncology Group (COG) cellbank

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newly Diagnosed Patients with ALL treated with Methotrexate
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2003-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Molecular basis for human reduced folate carrier (hRFC) transcripts | Up to 4 years
Correlation of hRFC expression and methotrexate transport and sensitivities | Up to 4 years
High frequency gene/transcript variants for hRFC in relation to response and resistance to methotrexate | Up to 4 years
Multidrug resistance-associated proteins in relation to response and resistance to methotrexate and mercaptopurine | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Larry Matherly, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States